CLINICAL TRIAL: NCT03353909
Title: The Efficacy of A New Crosslinked Hyaluronan Gel in the Prevention of Postoperative Intrauterine Adhesion After Dilatation and Curettage in Women With Delayed Miscarriage: A Prospective, Randomized, Controlled Trial
Brief Title: The Efficacy of A New Crosslinked Hyaluronan Gel in Prevention of Intrauterine Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioRegen Biomedical (CHangzhou) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FNL-2016-03
Record Dates: First submitted 2017-10-10; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Intrauterine Adhesion
Keywords: Intrauterine adhesion; Delayed miscarriage; hyaluronan gel
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): At the end of the dilatation and curettage, new crosslinked hyaluronan gel (3ml) was applied to the uterine cavity in women assigned to the treatment group through a 15-cm sterile cannula.
  Interventions: Device: new crosslinked hyaluronan gel
- Control (No Intervention): At the end of the dilatation and curettage, nothing was applied to the uterine cavity in women assigned to the control group.

INTERVENTIONS:
Device: new crosslinked hyaluronan gel — At the end of the dilatation and curettage, new crosslinked hyaluronan gel was applied to the uterine cavity.
  Other Names: MateRegen Gel
  Arms: Treatment

SUMMARY:
Using American Fertility Society classification of intrauterine adhesions, the efficacy of a new crosslinked hyaluronan gel in reducing intrauterine adhesion formation after dilatation and curettage for delayed miscarriage in women without previous dilatation and curettage was examined.

DETAILED DESCRIPTION:
Study Objectives: To evaluate the efficacy of a new crosslinked hyaluronan gel in reducing intrauterine adhesions formation after dilatation and curettage.

Design: Randomized controlled trial. Settings: Six hospitals for maternal and child health care in China. Patients: Three hundred women undergoing dilatation and curettage for delayed miscarriage without previous dilatation and curettage.

Interventions: Women were randomly assigned into either dilatation and curettage alone group or dilatation and curettage plus new crosslinked hyaluronan gel application group with 1:1 allocation.

Measurements and Outcomes: All patients were evaluated using American Fertility Society classification of IUAs during the follow-up diagnostic hysteroscopy, scheduled 3 months after dilatation and curettage procedure. The primary outcome was the number of women with IUAs, and the secondary outcome was the adhesion scores and the severity of IUAs.

ELIGIBILITY:
The inclusion criteria:

* Patients to be female, aged 18-45 years
* Without previous dilatation and curettage
* Undergoing dilatation and curettage for the current delayed miscarriage
* All participants should be with normal liver/rental function and without systemic disease
* Agree to use adequate forms of contraception throughout the study
* Be in good compliance with the follow-up examination according to the study protocol.

The exclusion criteria:

* Known/suspected intolerance or hypersensitivity to hyaluronan or its derivatives
* Genital tract malformation
* Inflammation of genital tract or pelvic cavity, clinical evidence of cancer in genital tract
* Suspected genital tuberculosis
* Abnormal blood coagulation
* Medical histories of peripheral vascular disease, alcohol/drug abuse, and mental illness
* Acute or severe infection
* Autoimmune diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of intrauterine adhesion | 3 months after dilatation and curettage
  The number of women with intrauterine adhesion

SECONDARY OUTCOMES:
The adhesion scores of extent of uterine cavity involved | 3 months after dilatation and curettage
  Evaluated according to American Fertility Society classification of intrauterine adhesion during the follow-up diagnostic hysteroscopy: 1 point (<1/3 cavity with adhesion), 2 points (1/3-2/3 cavity with adhesion) and 4 points (>2/3 cavity with adhesion), high values represent worse outcome
The adhesion scores of type of adhesion | 3 months after dilatation and curettage
  Evaluated according to American Fertility Society classification of intrauterine adhesion during the follow-up diagnostic hysteroscopy: 1 point (filmy adhesion), 2 points (filmy & dense adhesion) and 4 points (dense adhesion), high values represent worse outcome
The adhesion scores of menstrual pattern | 3 months after dilatation and curettage
  Evaluated according to American Fertility Society classification of intrauterine adhesion during the follow-up diagnostic hysteroscopy: 0 point (normal), 2 points (hypomenorrhea) and 4 points (amenorrhea), high values represent worse outcome
Cumulative adhesion score | 3 months after dilatation and curettage
  The summed score of the adhesion scores of extent of uterine cavity involved, type of adhesion and menstrual pattern; range: 1-12 points, high values represent worse outcome
Severity | 3 months after dilatation and curettage
  Graded according to cumulative adhesion score: Stage I (mild)(1-4 points), Stage II (moderate)(5-8 points) and Stage III (severe)(9-12 points).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Wu L, Zhou Y, Fan X, Huang J, Wu J, Yu R, Lou J, Yang M, Yao Z, Xue M. New Crosslinked Hyaluronan Gel for the Prevention of Intrauterine Adhesions after Dilation and Curettage in Patients with Delayed Miscarriage: A Prospective, Multicenter, Randomized, Controlled Trial. J Minim Invasive Gynecol. 2019 Jan;26(1):94-99. doi: 10.1016/j.jmig.2018.03.032. Epub 2018 Apr 17. PMID 29678756

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03353909/Prot_SAP_000.pdf